CLINICAL TRIAL: NCT05334355
Title: Impact of a Family History of Hypertension and Physical Activity on Left Ventricular Mass
Status: Completed | Type: Observational
Sponsor: Montclair State University (Other)
Responsible Party: Principal Investigator, Evan Matthews, Associate Professor, Montclair State University
Other Study IDs: IRB-FY15-16-185 & 19-20-1602
Record Dates: First submitted 2022-04-01; First posted 2022-04-19 (Actual); Results first posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Genetic Predisposition; Genetic Hypertension
MeSH Terms: conditions — Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Positive Family History of Hypertension: Young normotensive generally healthy adult with one or more biological parents with diagnosed hypertension.
  Interventions: Other: Family history of hypertension
- Negative Family History of Hypertension: Young normotensive generally healthy adult with no biological parent with diagnosed hypertension.

INTERVENTIONS:
Other: Family history of hypertension — Presence or absence of a family history of hypertension in a cross sectional study design.
  Groups: Positive Family History of Hypertension

SUMMARY:
This is a retrospective analysis of data collected within two previous studies. The data has been combined and used to investigate the impact of having a family history of hypertension on left ventricular muscle mass with and without controlling for moderate and vigorous intensity physical activity frequency per week. The hypothesis was that in a sample of mostly active participants, no differences in left ventricular mass between family history of hypertension groups would be observed, but the positive family history of hypertension group would have elevated left ventricular mass compared to the negative family history of hypertension group following statistical control of activity frequency.

DETAILED DESCRIPTION:
A positive family history of hypertension (FHH) (+FHH) is associated with elevated left ventricular mass (LVM). Regular physical activity (PA) may eliminate differences in LVM between +FHH and negative family history of hypertension (-FHH) adults. PURPOSE: To determine if a +FHH is associated with a greater LVM compared to a -FHH group within a sample of young, mostly active healthy adults with and without statistically controlling for PA. METHODS: Healthy young (18-32yrs) participants self-reported FHH status and habitual moderate and vigorous PA frequency. Participants then underwent an echocardiogram.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy

Exclusion Criteria:

* Known hypertension, cardiovascular disease, current pregnancy, current infectious disease, diabetes mellitus, kidney disease, a history of cancer, pulmonary disease, history of a stroke, obesity (for most people this means a body mass index greater than 30), or any life threatening chronic conditions

Ages: 18 Years to 32 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young healthy normotensive adults who are capable of self reporting family history of hypertension.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2016-04-19 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evan L Matthews, PhD, Principal Investigator — Montclair State University

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data is available on the Montclair State University Digital Commons website.
Time Frame: The data is currently available with no expiration date.
Access Criteria: Publicly available
URL: https://digitalcommons.montclair.edu/data/10

REFERENCES:
- [Result] Callaghan KN, Hosick PA, Brian MS, Matthews EL. Impact of a family history of hypertension and physical activity on left ventricular mass. J Sports Med Phys Fitness. 2023 Aug;63(8):949-956. doi: 10.23736/S0022-4707.23.14877-8. Epub 2023 May 9. PMID 37158799
- Available data/document: Individual Participant Data Set — https://digitalcommons.montclair.edu/data/10 — Complete individual participant data set is publicly available on the Montclair State University Digital Commons.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Positive Family History of Hypertension | Negative Family History of Hypertension
Started | 37 | 37
Completed | 29 | 32
Not Completed | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Positive Family History of Hypertension | Negative Family History of Hypertension | Total
Number analyzed (Participants) | 29 | 32 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 32 | 61
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.44827586 (2.384266987) | 22.6875 (2.966887149) | 23.04918033 (2.7106)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 37
  Male | 11 | 13 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 8 | 12
  Not Hispanic or Latino | 25 | 24 | 49
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29 | 32 | 61
Left Ventricular Mass/Body Surface Area [Mean (Standard Deviation); unit: grams/meter squared] | 88.35017813 (17.30587475) | 73.51184729 (17.74896472) | 80.56613572 (18.9302)

OUTCOME MEASURES:

1. Primary Outcome: Left Ventricular Mass
Description: Muscle mass in grams of the left ventricle of the heart as estimated by ultrasound.
Time Frame: Day 2
Measure: Mean (Standard Deviation); unit: gram
Arm/Group | Positive Family History of Hypertension | Negative Family History of Hypertension
Number analyzed (Participants) | 29 | 32
gram | 155.1680523 (42.6141251) | 129.5013331 (41.76454204)

ADVERSE EVENTS:
Time Frame: 3 years, 10 months
Description: There were no adverse events or mortality in this study. This was an observational cross-sectional study with no intervention.
Arm/Group | Positive Family History of Hypertension | Negative Family History of Hypertension
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/32
Other Adverse Events (participants affected / at risk) | 0/29 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-14): https://cdn.clinicaltrials.gov/large-docs/55/NCT05334355/Prot_SAP_000.pdf